CLINICAL TRIAL: NCT06175650
Title: Towards a Sex-specific "Female Enhanced Recovery After Cardiac Surgery'' (F-ERAS) Pathway: An Observational Registration and Evaluation of Characteristics and Perioperative Management of Cardiac Surgery Patients
Brief Title: Towards a Sex-specific "Female Enhanced Recovery After Cardiac Surgery'' (F-ERAS) Pathway:
Acronym: F-ERAS
Status: Recruiting | Type: Observational
Sponsor: Jennifer Breel (Other)
Responsible Party: Sponsor-Investigator, Jennifer Breel, Investigator, Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: W22_051 # 22.082
Record Dates: First submitted 2022-03-20; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Female; Male; Surgery,Cardiac
Keywords: Anesthesia; Quality of Life
MeSH Terms: interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female: Female patients undergoing cardiac surgery
  Interventions: Procedure: Cardiac surgery
- Male: Male patients undergoing cardiac surgery
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Cardiac surgery of all types

SUMMARY:
The aim of this study is to evaluate the differences between men and women undergoing cardiac surgery. We will look at perioperative factors such as body weight, body surface area, previous medical history, pharmacokinetics, transfusion, coagulation, cardiopulmonary bypass (CPB) related factors, cardiac function, inotropic requirements, risk, and outcome scores as well as morbidity and mortality at 30 and 90 days, 1, 5, and 10 years.

DETAILED DESCRIPTION:
Observational, multicentre, retrospective data collection from the mandatory Quality Assurance database (the Netherlands Heart Registry, (NHR), supplemented with data from the electronic patient files (EPIC). The retrospective data is already available.

In addition, we will continue the retrospective study into a prospective registry of data after the analysis of the retrospective data. Patients will be approached one, five and ten years after the operation and a questionnaire will be sent to document quality of life. No research-related interventions other than questionnaires will be performed

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years
* All patients who underwent cardiac surgery from 1 January 2016 to the start of the study, in either of the centres (AMC or VUmc) (retrospective)
* All patients undergoing cardiac surgery from the start of the study (~March 2022) until approximately 2032

Exclusion Criteria:

• Patients who object to the re-use of their care data or do not give consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female patients, 18 years and older. The study group consists of all patients who underwent cardiac surgery from 1 January 2016 onwards, in either of the centres (AMC or VUmc). The registry will continue for at least 10 years after the inclusion of the last patient.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-11-21 (Estimated); Study Completion 2026-11-21 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | up to 30 days post-surgery
  Incidence of mortality (number of patients) specific (coagulation), transfusion products, anesthesia, surgery and cross-clamp times, etc
Primary endpoint | up to 30 days post-surgery
  incidence of cerebrovascualar accident with neurological sequelae (number of patients)
Primary endpoint | up to 30 days post-surgery
  incidence of acute kidney injury (number of patients)
Primary endpoint | up to 30 days post-surgery
  incidence of low cardiac output syndrome, pulmonary and other complications (requiring ventilation > 48 hours post-operatively)
Primary endpoint | up to 30 days post-surgery
  Number of specific (coagulation), transfusion products,
Primary outcome | up to 30 days post-surgery or if still in hospital, until discharge
  Times: surgical, cross-clamp, bypass, anesthetic, intensive care admission, hospital admission, etc.

SECONDARY OUTCOMES:
Morbidity and mortality | At 30, 90, 365 days
  peroperative and post-operative complications
Survival | At 5 and 10 years
  Long term survival
Health related Quality of life measured by PROMS | At 1, 5 and 10 years
  Long term quality of life after cardiac surgery, measured by Seattle Angina Questionaire (SAQ), EuroQol Quality of life (EQ-5D-5L) and Coronary Revascularisation Outcome Questionnaire (CROQ) or other appropriate questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Hollmann, Professor, Principal Investigator — Anesthesiology and Pain Medicine, Amsterdam Medical Center
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cho L, Kibbe MR, Bakaeen F, Aggarwal NR, Davis MB, Karmalou T, Lawton JS, Ouzounian M, Preventza O, Russo AM, Shroyer AW, Zwischenberger BA, Lindley KJ. Cardiac Surgery in Women in the Current Era: What Are the Gaps in Care? Circulation. 2021 Oct 5;144(14):1172-1185. doi: 10.1161/CIRCULATIONAHA.121.056025. Epub 2021 Oct 4. PMID 34606298
- [Background] Dixon LK, Di Tommaso E, Dimagli A, Sinha S, Sandhu M, Benedetto U, Angelini GD. Impact of sex on outcomes after cardiac surgery: A systematic review and meta-analysis. Int J Cardiol. 2021 Nov 15;343:27-34. doi: 10.1016/j.ijcard.2021.09.011. Epub 2021 Sep 11. PMID 34520795
- [Background] Nanegrungsunk D, Patel S, Jan T, Ngai JY. Preoperative Care Practice for Female Cardiac Patients: A Survey From the Society of Cardiovascular Anesthesiologists. J Cardiothorac Vasc Anesth. 2022 Mar;36(3):920-921. doi: 10.1053/j.jvca.2021.09.054. Epub 2021 Oct 3. No abstract available. PMID 34776353
- [Background] Peters SAE, Kluin J. Why do women do worse after coronary artery bypass grafting? Eur Heart J. 2021 Dec 28;43(1):29-31. doi: 10.1093/eurheartj/ehab617. No abstract available. PMID 34524421